CLINICAL TRIAL: NCT05748977
Title: Inhaled Fenotereol,Ipratroium Plus Beclomethasone Versus Salmeterol,Tiotropium Plus Fluticasone in Frequent Excerbator COPD Patients
Brief Title: Short Acting Agents Vs Long Acting in Frequent Excerbator COPD Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nermen Abuelkassem, lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SABA,SAMA versus LABA,LAMAcopd
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Copd
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SABA,SAMA ICS (Experimental)
  Interventions: Drug: SABA SAMA ICS Vs LABA LAMA ICs
- LABA,LAMA ICS (Experimental)
  Interventions: Drug: SABA SAMA ICS Vs LABA LAMA ICs

INTERVENTIONS:
Drug: SABA SAMA ICS Vs LABA LAMA ICs — Short acting agents,long acting agents ,ics

SUMMARY:
Chronic obstructive pulmonary disease is heterogeneous lung condition characterized by chronic respiratory symptoms (dyspnea, cough, sputum production, exacerbations) due to abnormalities of the airways (bronchitis, bronchiolitis) and/or alveoli (emphysema) that cause persistent, often progressive ,airflow obstruction.

There are network meta analysis to compare the efficacy and safety of short acting bronchodilators Vs long acting agents in treatment of COPD

DETAILED DESCRIPTION:
Aim of the work1.To compare efficacy of short acting beta 2 agonists ,short acting antimuscrinic agents and beclomethasone versus long acting beta 2 agonist,short acting antimuscurnic agents and fluticasone.- Type of the study: This study is a randomized controlled trail 2.4. 2- Study Setting: Present study will be conducted in chest outpatient clinic Chest department Assiut University hospital 2.4. 3- Study subjects: Frequent exacerbator COPD patients Based on determining the main outcome variable, the estimated minimum required sample size is 80 patients (40 in each group).

Main outcome variable is difference in dyspnoea scores in frequent exacerbator COPD patients receiving long-acting steroids vs. short acting treatment. Based on previous systematic review we expected to find significant improvement in long-acting treatment group (large effect size). Data will be collected through: patients diagnosed COPD by different investigations (history, examinations spirometry) have recurrent exacerbations, some patients receiving short acting beta 2 agonists, short acting anti-muscurnic agents and beclomethasone versus long acting agents and fluticasone then all patients followed using dyspnea scores, CCQ, saint George questionnaire which assess heath related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* All frequent exacerabator copd patients

Exclusion Criteria:

* patients less than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-20 (Estimated); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-03-20 (Estimated)

PRIMARY OUTCOMES:
to assess improvement of symptoms mainly dyspnea | 1 year
  to assess dyspnea in two groups by mMRC,saint gorge quetsonaire

CONTACTS AND LOCATIONS:
Overall Officials: nermen M abuelkassem, Lecturer, Principal Investigator — MD
Locations (1):
- Nermen Mohammed Abuelkassem, Asyut, Egypt